CLINICAL TRIAL: NCT05093179
Title: The Effect of Deep Tissue Massage on Respiratory Parameters in Healthy People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Bartosz Trybulec, Assistant professor, Jagiellonian University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1072.6120.7.2019
Record Dates: First submitted 2021-09-30; First posted 2021-10-26 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Spirometry; Massage
Keywords: deep tissue; massage; spirometry; chest; fascial release

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deep tissue massage group (Experimental): The one session of deep tissue massage was performed. The patient's positions were changed depending on the specificity of used techniques.
  The following techniques were used:
  * Shifting the rectus abdominis m.,
  * Stretching of the fascia within the costal arches,
  * trigger points compression (30-60 s).
  * Stretching of the chest fascia, superficially with forearm or fingertips on intercostal muscles,
  * "filleting" the pectoral muscles,
  * "hook and stretch" with the proximal phalanges of the fingers 2-4 and the forearm
  * "filleting" between the pectoral muscles and the deltoids,
  * Releasing the lateral edge of the scapula using the fingers and stretching the tissues, Releasing the medial edge of the scapula using the fingers and the weight of the patient,
  * "hook and stretch" of the trapezius muscle,
  * Subsequently, the patient took a prone position.
  * Stretching of the levator scapulae and supraspinatus muscles using the fist, forearm and elbow were performed.
  Interventions: Procedure: Deep tissue massage
- Classic massage group (Active Comparator): The one session of classic massage was performed. The massage was performed with moderate force. The entire procedure took about 15-20 min. The sequence of standard classic massage techniques was used in standard way and patterns.
  Interventions: Procedure: Classic massage

INTERVENTIONS:
Procedure: Deep tissue massage — Administered as a soft tissue mobilization performed by the therapist with fingertips, knuckles, elbows and/or fists on the tissues that manifest symptoms of fascial restrictions. The techniques were performed with individually adjusted force until the change (eg. increased mobility) in the tissue being treated was stated by the therapist.
  Arms: Deep tissue massage group
Procedure: Classic massage — The subject was lying supine on the table, with a roller placed under the knee joints, the upper limbs along the body. The following sequence of techniques was used in the longitudinal and transverse strands and in the intercostal spaces (excluding the breast in women): effleurage, friction, petrissage, pressures, tapotement and vibrations.
  Arms: Classic massage group

SUMMARY:
Deep tissue massage (DTM), based on deep palpation and elimination of fascia restrictions, can reduce symptoms resulting from fascial disorders. The goal of this study was the analysis of the DTM effect on respiratory parameters in healthy people. People of both sexes living in the city of Cracow were recruited to the study by the authors personally and through social media. An original questionnaire was completed in the presence of the examiner in order to collect the participants characteristics data. Questions about past diseases, previous surgical procedures or injuries, currently taken medications or the level of physical activity were asked to check the inclusion/exclusion criteria. The study involved a group of 40 people divided into two subgroups. The experimental group underwent a single DTM session. Classic massage was performed in the control group. Before and after treatment the lung vital capacity, chest circumference and oxygen saturation were measured and a spirometry test was performed. The main hypothesis assumed that static respiratory parameters should increase after the treatment session more in the experimental than in control group while the dynamic respiratory parameters would not differ significantly in both groups before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Physical activity of minimum 30 min. duration, at least 3 times a week.
2. No chest injuries.
3. No contraindications for DTM/classic massage.
4. No serious diseases of the respiratory and/or cardiovascular systems.
5. No tobacco products smoking (incl.e-smoking).
6. No posture defects that could affect the chest mobility.

Exclusion Criteria:

1. Contraindications to DTM/classic massage of the chest.
2. Occurrence of serious diseases of the respiratory/cardiovascular system now or in the past.
3. Lack of or low physical activity (< 30 min min. 3 times per week).
4. Tobacco smoking (incl.e-smoking).
5. Chest injuries.
6. Posture defects that may affect the chest mobility.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Assessment of change of lung vital capacity | twice: before and immediately after procedure administration in both groups
  The vital capacity of the lungs was assessed with spirotest (Riester, mod. 5260). The subject stood with legs hip-width apart. For each measurement, disposable cardboard mouthpieces were used. The examined person held the device vertically with both hands. At the examiner's command, subject took in as much air as possible, then tightly bit the mouthpiece with his mouth, and with all of their strength, exhaled air into the device for as long as possible. The subject had only 1 attempt-measured values were recorded with an accuracy of 50 mL.
Assessment of change of blood oxygen saturation | twice: before and immediately after procedure administration in both groups
  Testing blood oxygen saturation was performed in a sitting position with digital pulseoximeter CMS50D. The device was put on the second finger of the left hand each time. The highest value displayed by the pulseoximeter within 30 s was recorded with an accuracy of 1%.
Assessment of change of chest circumference | twice: before and immediately after procedure administration in both groups
  The chest circumference was measured with a measuring tape, wrapped horizontally around the chest at the level of the xiphoid process. The subject was standing with feet hip-width apart, arms hanging along the body. At the command, the subject would take a maximum breathe in (first measurement) and exhale to the maximum for the next (second measurement). Obtained values were recorded with an accuracy of 0.5 cm.
Asessment of change of Peak Expiratory Flow | twice: before and immediately after procedure administration in both groups
  Dynamic spirometry test was performed, assessing the peak expiratory flow (PEF) measured in liters per second [l/s]. The test was performed with PNEUMO® spirometer and PNEUMO 2005 software (abcMED). The subject was sitting with his legs on the floor-hip joint flexed at an angle of 70o-90o and carried out the following command: "Breathe calmly. On my command, breathe in as much as possible, as quickly as possible, as intensively as possible, and while at the top of the inhalation, without waiting, breathe out as hard and as long as possible ". This cycle was performed at least 3 times obtaining 3 measurements according to the standard ERSATS 2005.
Assessment of change of Peak Inspiratory Flow | twice: before and immediately after procedure administration in both groups
  Dynamic spirometry test was performed, assessing the peak inspiratory flow (PIF) measured in liters per second [l/s]. The test was performed with PNEUMO® spirometer and PNEUMO 2005 software (abcMED). The subject was sitting with his legs on the floor-hip joint flexed at an angle of 70o-90o and carried out the following command: "Breathe calmly. On my command, breathe in as much as possible, as quickly as possible, as intensively as possible, and while at the top of the inhalation, without waiting, breathe out as hard and as long as possible ". This cycle was performed at least 3 times obtaining 3 measurements according to the standard ERSATS 2005.
Assessment of change of Forced Vital Capacity | twice: before and immediately after procedure administration in both groups
  Dynamic spirometry test was performed, assessing the forced vital capacity (FVC), measured in liters. The test was performed with PNEUMO® spirometer and PNEUMO 2005 software (abcMED). The subject was sitting with his legs on the floor-hip joint flexed at an angle of 70o-90o and carried out the following command: "Breathe calmly. On my command, breathe in as much as possible, as quickly as possible, as intensively as possible, and while at the top of the inhalation, without waiting, breathe out as hard and as long as possible ".
Assessment of change of Maximum Expiratory Flow. | twice: before and immediately after procedure administration in both groups
  Dynamic spirometry test was performed, assessing the maximum expiratory flow (MEF), measured in liters per second. The test was performed with PNEUMO® spirometer and PNEUMO 2005 software (abcMED). The subject was sitting with his legs on the floor-hip joint flexed at an angle of 70o-90o and carried out the following command: "Breathe calmly. On my command, breathe in as much as possible, as quickly as possible, as intensively as possible, and while at the top of the inhalation, without waiting, breathe out as hard and as long as possible ". This cycle was performed at least 3 times obtaining 3 measurements according to the standard ERSATS 2005.
Assessment of change of Forced Expiratory Volume | twice: before and immediately after procedure administration in both groups
  Dynamic spirometry test was performed, assessing the forced expiratory volume in 1 s (FEV1) measured in liters. The test was performed with PNEUMO® spirometer and PNEUMO 2005 software (abcMED). The subject was sitting with his legs on the floor-hip joint flexed at an angle of 70o-90o and carried out the following command: "Breathe calmly. On my command, breathe in as much as possible, as quickly as possible, as intensively as possible, and while at the top of the inhalation, without waiting, breathe out as hard and as long as possible ". This cycle was performed at least 3 times obtaining 3 measurements according to the standard ERSATS 2005.
Assessment of change of Maximum Voluntary Ventilation | twice: before and immediately after procedure administration in both groups
  Dynamic spirometry test was performed, assessing the maximum voluntary ventilation (MVV) measured in liters per minute. The test was performed with PNEUMO® spirometer and PNEUMO 2005 software (abcMED). The subject was sitting with his legs on the floor-hip joint flexed at an angle of 70o-90o and carried out the following command: "Breathe calmly. On my command, inhale and exhale as quickly and as deeply as possible for 15 s until you hear the 'stop' command. This cycle was performed at least 3 times obtaining 3 measurements according to the standard ERSATS 2005.

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz T. trybulec, PhD, Study Director — Jagiellonian University Medical College in Cracow
Locations (1):
- Institute of Physiotherapy Jagiellonian University Medical College, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No